CLINICAL TRIAL: NCT03317964
Title: Genetic Basis of Pacing-Induced Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1706-34
Record Dates: First submitted 2017-10-16; First posted 2017-10-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pacemaker, Artificial; Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saliva - cardiomyopathy: Saliva sample for genetic testing from subjects who developed cardiomyopathy
  Interventions: Other: Saliva sample
- Saliva - no cardiomyopathy: Saliva sample for genetic testing from subjects who do not have cariomyopathy
  Interventions: Other: Saliva sample

INTERVENTIONS:
Other: Saliva sample — Extract sample of saliva only once

SUMMARY:
The purpose of this study is to collect a saliva sample from patients with a pacemaker to study genes involved in cardiomyopathy, a condition where the heart muscle is abnormal.

DETAILED DESCRIPTION:
DNA will be extracted from the saliva to test for changes in genes related to cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been assessed for cardiomyopathy

Exclusion Criteria:

* Patients who do not have adequate follow up care to determine if they do or do not have cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Robert Packer Hospital, Sayre, PA
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with genotype frequency | through study completion, an average of 1 year
  Number of participants with genotype frequency based on genetic testing of saliva samples

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Deshmukh, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No